CLINICAL TRIAL: NCT00001893
Title: A Clinical Trial of TNFR:Fc in a Segmental Allergen Challenge Model of Asthma
Brief Title: Study of TNFR:Fc (Enbrel) in the Treatment of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Steward Levine, M.D./National Heart, Lung and Blood Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 990140; 99-H-0140
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-13

CONDITIONS: Asthma
Keywords: Bronchoprovocation; Airway Inflammation; Tumor Necrosis Factor; Bronchoalveolar Lavage; Pulmonary Function Test; Asthma
MeSH Terms: conditions — Asthma | interventions — Etanercept

INTERVENTIONS:
Drug: TNFR:Fc

SUMMARY:
The proposed study is a phase II clinical trial of TNFR:Fc therapy in a segmental allergen bronchoprovocation model of atopic asthma. The goal of this study is to assess whether inhibition of tumor necrosis factor (TNF) bioactivity can attenuate airway inflammation in mild-to-moderate allergic asthmatics. This protocol will utilize a randomized, double-blind, placebo-controlled trial design. TNF bioactivity will be inhibited via systemic administration (e.g., subcutaneous injection) of a dimeric fusion protein consisting of the extracellular ligand binding domain of the 75-kilodalton TNF receptor linked to the Fc portion of human IgG1 (TNFR:Fc, Immunex). The data generated by this study will address the utility of anti-TNF therapy for patients with asthma.

DETAILED DESCRIPTION:
The proposed study is a phase II clinical trial of TNFR:Fc therapy in a segmental allergen bronchoprovocation model of atopic asthma. The goal of this study is to assess whether inhibition of tumor necrosis factor (TNF) bioactivity can attenuate airway inflammation in mild-to-moderate allergic asthmatics. This protocol will utilize a randomized, double-blind, placebo-controlled trial design. TNF bioactivity will be inhibited via systemic administration (e.g., subcutaneous injection) of a dimeric fusion protein consisting of the extracellular ligand- binding domain of the 75-kilodalton TNF receptor linked to the Fc portion of human IgG1 (TNFR:Fc, Immunex). The data generated by this study will address the utility of anti-TNF therapy for patients with asthma.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be between 18 and 65 years of age, male or female, and must be at least 5 feet in height.

The diagnosis of asthma requires a history of intermittent, reversible expiratory flow limitation.

Patients will have mild-to-moderate allergic asthma as defined by a baseline forced expiratory flow in one second (FEV(1)) greater than 70% of predicted (at least 6 hours after bronchodilator use) and therapy limited to inhaled beta-agonists.

Patients must be without evidence of an asthma exacerbation or a viral upper respiratory tract infection for 6 weeks prior to entry into the study.

Positive skin prick-puncture test to one or more common aeroallergens.

A positive inhaled methacholine challenge as defined by a decrease in FEV(1) of at least 20% (PC20) in response to inhalation of less than 25 mg/ml of methacholine.

A decrease in FEV(1) of at least 20% in response to inhalation of up to 10,000 bioequivalency allergy units (BAU) or allergy units (AU) per ml of a selected common aeroallergen (house dust mite, cat hair or grasses) or up to 150 Antigen E units per ml of short ragweed. Asthmatic patients must also demonstrate a late asthmatic response (defined as a 20% fall from the baseline established following completion of the early asthmatic response).

Normal complete blood count, PT, PTT, and serum electrolytes, mineral and hepatic panels (less than 30 ml of blood will be drawn), normal EKG and chest radiograph without acute pulmonary infiltrates.

For women of childbearing potential, negative pregnancy test with 2 weeks prior to study and willingness to adhere to reliable birth control methods during the study.

EXCLUSION CRITERIA:

Hypersensitivity to TNFR:Fc

Women who are breast-feeding infants will be excluded because the risk of a serious adverse reaction in the infants to TNFR:Fc is unknown.

Diagnosis of a pulmonary disorder other than asthma (e.g., chronic bronchitis, cystic fibrosis, bronchiectasis, HIV-related lymphocytic airway inflammation).

Respiratory tract infection or asthma exacerbation within 4 weeks of screening.

Presence of an active infection.

Use of theophylline, oral or inhaled corticosteroid, nedocromil sodium, cromolyn sodium, zilueton, leukotriene receptor antagonists (e.g., zafirlukast or montelukast), or anti-cholinergic agents within the prior 3 months. In addition, patients requiring ongoing therapy with anti-histamines, hydroxyzine, and tricyclic anti-depressants will be excluded. Research subjects can continue therapy with inhaled beta-agonists during the study.

History of anaphylaxis or severe allergic response.

History of adverse reactions to lidocaine or other local anesthetics.

Use of aspirin within 2 weeks of the bronchoscopic study or non-steroidal anti-inflammatory agents within 2 days of the bronchoscopic study.

History of cigarette smoking within the past 3 years.

History of allergy immunotherapy within the past year.

Allergy to methacholine.

Positive test for human immunodeficiency virus (to exclude patients with HIV-related lymphocytic airway inflammation).

Positive test for hepatitis viruses (to exclude patients with hepatitis-related lung disease, such as pleural effusions, interstitial pneumonitis and fibrosis).

History of Crohn's disease (to exclude patients with inflammatory bowel disease-related alveolar lymphocytosis).

History of diseases associated with impaired host defenses, such as diabetes mellitus or congestive heart failure. Patients with impaired host defenses also include individuals with either acquired or congenital, quantitative or qualitative defects in neutrophil, lymphocyte, monocyte/macrophage or complement function. Similarly, patients requiring immunosuppressive therapies, such as a chronic corticosteroid utilization for more than 6 months or cytoxic chemotherapeutic agents will be excluded.

History of chronic heart failure or coronary artery disease.

History of central nervous system demyelinating disorders, such as multiple sclerosis, myelitis or optic neuritis.

History of hematologic disorders, such as anemia (other than iron deficiency anemia), thrombocytopenia or leukopenia.

History of renal disease, such as chronic renal failure or renal artery stenosis with renal artery stent placement.

History of psoriasis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1999-08-17; Primary Completion 2002-12-31 (Actual)

PRIMARY OUTCOMES:
Whether subcutaneous administration of TNFR:Fc alters TNF bioactivity in brochoalveolar lavage fluid (BALF) samples. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Broide DH, Lotz M, Cuomo AJ, Coburn DA, Federman EC, Wasserman SI. Cytokines in symptomatic asthma airways. J Allergy Clin Immunol. 1992 May;89(5):958-67. doi: 10.1016/0091-6749(92)90218-q. PMID 1374772